CLINICAL TRIAL: NCT05580692
Title: A Multinational, Multi-center, Prospective Cohort Study Evaluating Seroprevalence and Seroconversion of Antibodies Against Adeno-associated Virus (AAV) Serotypes in Subjects With Hemophilia A
Brief Title: A Prospective Study Evaluating Seroprevalence and Seroconversion of Antibodies Against Adeno-associated Virus (AAV)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision to terminate; sufficient sample size for statistical analysis has been achieved.
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 270-702
Record Dates: First submitted 2022-09-16; First posted 2022-10-14 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient Cohort (Experimental): All Patients are within the same arm
  Interventions: Procedure: Biospecimen Collection

INTERVENTIONS:
Procedure: Biospecimen Collection — Biospecimen Sample Collection

SUMMARY:
A prospective cohort study utilizing biospecimen sample collection from adult Hemophilia A subjects to evaluate and characterize seroprevalence and the seroconversion of antibodies against AAV serotypes

DETAILED DESCRIPTION:
This is a multinational, multi-center, prospective cohort study utilizing biospecimen sample collection from adult Hemophilia A subjects to evaluate and characterize seroprevalence and the seroconversion of antibodies against AAV serotypes

ELIGIBILITY:
Inclusion Criteria:

* Adult Subjects with Hemophilia A

Exclusion Criteria:

* Subject previously treated with AAV vector gene therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2023-03-14 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
To qunatify Seroprevalence of antibodies to selected AAV serotypes | 52 weeks
  Number of patients with detectable antibodies to selected AAV serotypes

SECONDARY OUTCOMES:
To describe and characterize selected AAV serotypes antibody responses in adult subjects with Hemophilia A | 52 weeks
  Antibody titer levels measured in target population to selected AAV serotypes

CONTACTS AND LOCATIONS:
Overall Officials: Medinfo Medinfo, Study Director — BioMarin Pharmaceutical
Locations (18):
- Argentina (4):
  - Instituto Hematologia Arbesu, Godoy Cruz, Mendoza Province
  - Hospital Ramon Jose Vidal, Corrientes
  - Medico Hematologo, Mendoza
  - Instituto de Hematologia y Medicina Clinica Dr. RUben Davoli, Rosario
- Australia (2):
  - Royal Prince Alfred Hospital, Camperdown
  - Haemophilia and Haemostasis Centre Level 1 Cancer Centre South Metropolitan Health Service Fiona Stanley Hospital, Murdoch
- Medical University of Vienna, Vienna, Austria
- Saudi Arabia (2):
  - King Faisal Specialist Hospital & Research Center, Riyadh
  - King Saud University Medical City King Saud University, Riyadh
- Sweden (2):
  - Skane University Hospital, Malmo
  - ME Centrum för kliniska cancerstudier - House H3, Solna
- Turkey (Türkiye) (6):
  - Acibadem Adana Hospital, Adana
  - Hacettepe University, Ankara
  - Gaziantep University Medical Faculty Sahinbey Educational Research Hospital, Gaziantep
  - Istanbul University Cerrahpasa - Cerrahpasa Medical Faculty, Istanbul
  - Ege University Medical Faculty, Izmir
  - Ondokuz Mayis Univ. Med. Fac., Samsun
- Sheikh Shakhbout Medical City, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No